CLINICAL TRIAL: NCT02044419
Title: A Phase 1, Open-label, Randomised, Crossover Study to Determine the Comparative Bioavailability of 20 mg Lomitapide Where the Contents Have Been Opened and Sprinkled in Applesauce or Mashed Banana ("Sprinkled Contents") to a Single Oral Capsule Dose of 20 mg Lomitapide ("Intact Capsule") in Healthy Subjects
Brief Title: A Comparative Bioavailability Study of Lomitapide 20 mg Intact vs Sprinkled
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AEGR-733-032
Record Dates: First submitted 2013-11-06; First posted 2014-01-24 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: Comparative; Bioavailability; lomitapide
MeSH Terms: interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- lomitapide sprinkled in applesauce (Experimental): Contents of single 20 mg capsule of lomitapide sprinkled in applesauce
  Interventions: Drug: lomitapide
- lomitapide sprinkled in mashed banana (Experimental): Contents of single 20 mg capsule of lomitapide sprinkled in mashed banana
  Interventions: Drug: lomitapide
- lomitapide (intact) (Experimental): Intact capsule of 20 mg lomitapide
  Interventions: Drug: lomitapide

INTERVENTIONS:
Drug: lomitapide
  Other Names: Juxtapid; Lojuxta

SUMMARY:
To compare the relative bioavailability of lomitapide when administered by sprinkling the contents of a 20 mg capsule of lomitapide in applesauce or in mashed banana to a single oral intact capsule dose of 20 mg lomitapide in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a non-smoking healthy male or female, aged between 18 and 40 years of age.
2. Subject has a BMI of 18.5 - 25 kg/m2.
3. Subject has total body weight between > 50 kg to ≤ 100 kg.
4. Subjects must agree to use acceptable methods of contraception.
5. All females, regardless of childbearing potential, must have a negative serum beta human chorionic gonadotropin pregnancy test at Screening and on admission.
6. In good health, determined by no clinically significant or relevant abnormalities identified by a detailed medical history & full physical examination.
7. No known history of hypersensitivity or previous intolerance to lomitapide, applesauce, and/or banana.
8. Subjects must be capable of understanding and complying with the requirements of the protocol and must have signed the informed consent form prior to undergoing any study-related procedures.

Exclusion Criteria:

1. Subject has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion.
2. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs.
3. Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations.
4. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;
5. Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) such as a QTcF interval of >450 msec, a history of a prolonged QTc interval or Brugada syndrome.
6. History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, allergic, dermatological, metabolic, neurological, psychiatric or other disease.
7. History or laboratory evidence of Gilbert's syndrome.
8. Positive results in any of the serology tests for Hepatitis B Surface Antigen (HbsAg), anti-Hepatitis core antibody (anti-HBc Ig G [and anti-HBc IgM if IgG is positive], Hepatitis C antibodies (anti-HCV), and HIV 1 and 2 antibodies, (anti-HIV 1/2).
9. Use of any drugs of abuse within 6 months prior to admission.
10. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates and methadone) or from the alcohol breath test at screening and on admission (Day -1).
11. History or clinical evidence of alcohol or drug abuse within one year prior to admission.
12. Mentally handicapped.
13. Participation in a drug trial within 90 days prior to first drug administration.
14. Use of any prescription medication within 2 weeks prior to admission (Day -1), with the exception of the oral contraceptive pill.
15. Use of any substance inducing or inhibiting CYP3A4 enzymes within 30 days prior to admission (Day -1).
16. Use of any over-the-counter (OTC) medication (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to admission (Day -1), unless deemed acceptable by the Investigator and Sponsor.
17. Use of alcohol-, grapefruit-, starfruit-, or caffeine-containing foods or beverages within 72 hours prior to admission and through Study Completion.
18. Donation of more than 500 mL of blood within 90 days prior to drug administration.
19. Receipt of blood products within 2 months prior to admission.
20. Poor peripheral venous access.
21. Use of any tobacco- or nicotine-containing products within 6 months prior to admission (Day -1).
22. Any acute or chronic condition, scheduled hospitalisation (inclusive of elective surgery during study), or scheduled travel prior to completion of all study procedures.
23. Any circumstances or conditions, which, in the opinion of the PI, may affect full participation in the trial or compliance with the protocol.
24. Legal incapacity or limited legal capacity at screening.
25. Subjects who are vegetarians, vegans or have any dietary restrictions conflicting with the study standardised menus.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2013-12-23 (Actual); Study Completion 2013-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sumeray, MD, Study Chair — Aegerion Pharmaceuticals, Inc.; Ulrike Lorch, MD, Principal Investigator — Richmond Phamacology, LTD
Locations (1):
- Richmond Pharmacology Ltd, Croydon, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Applesauce, Mashed Banana, Intact Capsule (ABC); Intact Capsule, Applesauce, Mashed Banana (CAB): First Intervention: Contents of single 20 mg capsule of lomitapide sprinkled in applesauce Second Intervention: Contents of single 20 mg capsule of lomitapide sprinkled in mashed banana Third Intervention: Intact capsule of 20 mg lomitapide
- Mashed Banana, Intact Capsule, Applesauce (BCA): First Intervention: Contents of single 20 mg capsule of lomitapide sprinkled in mashed banana Second Intervention: Intact capsule of 20 mg lomitapide Third Intervention: Contents of single 20 mg capsule of lomitapide sprinkled in applesauce
Period: First Intervention
Arm/Group | Applesauce, Mashed Banana, Intact Capsule (ABC) | Mashed Banana, Intact Capsule, Applesauce (BCA) | Intact Capsule, Applesauce, Mashed Banana (CAB)
Started | 11 | 10 | 11
Completed | 11 | 9 | 10
Not Completed | 0 | 1 | 1
Period: Second Intervention
Arm/Group | Applesauce, Mashed Banana, Intact Capsule (ABC) | Mashed Banana, Intact Capsule, Applesauce (BCA) | Intact Capsule, Applesauce, Mashed Banana (CAB)
Started | 11 | 9 | 10
Completed | 11 | 9 | 10
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Applesauce, Mashed Banana, Intact Capsule (ABC) | Mashed Banana, Intact Capsule, Applesauce (BCA) | Intact Capsule, Applesauce, Mashed Banana (CAB)
Started | 11 | 9 | 10
Completed | 11 | 9 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Applesauce, Mashed Banana, Intact Capsule (ABC): Contents of single 20 mg capsule of lomitapide sprinkled in applesauce, mashed banana
  Capsule taken intact
  lomitapide
- Mashed Banana, Intact Capsule, Applesauce (BCA); Intact Capsule, Applesauce, Mashed Banana (CAB): Contents of single 20 mg capsule of lomitapide sprinkled in applesauce& mashed banana
  Capsule taken intact
  lomitapide
- Total: Total of all reporting groups
Arm/Group | Applesauce, Mashed Banana, Intact Capsule (ABC) | Mashed Banana, Intact Capsule, Applesauce (BCA) | Intact Capsule, Applesauce, Mashed Banana (CAB) | Total
Number analyzed (Participants) | 11 | 10 | 11 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 11 | 32
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.45 (5.837) | 25.90 (5.131) | 27.91 (3.27) | 27.42 (4.746)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 6 | 15
  Male | 8 | 4 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 10 | 10 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 4 | 9
  White | 7 | 6 | 5 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 10 | 11 | 32

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t
Description: Area under the concentration-time curve from hour 0 to the last measurable concentration of lomitapide and its metabolites (M1& M3).
Time Frame: predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Population: Pharmacokinetic Analysis Set included all subjects who received at least one single dose of lomitapide and who had evaluable PK data
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Lomitapide Sprinkled in Applesauce (Treatment A): Contents of single 20 mg capsule of lomitapide sprinkled in applesauce
- Lomitapide Sprinkled in Mashed Banana (Treatment B): Contents of single 20 mg capsule of lomitapide sprinkled in mashed banana
- Intact Capsule of 20 mg Lomitapide (Treatment C): Intact capsule of 20 mg lomitapide
Arm/Group | Lomitapide Sprinkled in Applesauce (Treatment A) | Lomitapide Sprinkled in Mashed Banana (Treatment B) | Intact Capsule of 20 mg Lomitapide (Treatment C)
Number analyzed (Participants) | 30 | 30 | 30
ng*h/mL
  Lomitapide | 38.3 (15.2) | 40.2 (13.4) | 43.6 (17.7)
  M1 | 70.4 (20.2) | 72.9 (23.1) | 75.2 (22.8)
  M3 | 443 (308) | 450 (292) | 460 (325)

2. Primary Outcome: Cmax
Description: Maximum observed concentration of lomitapide and its metabolites (M1& M3).
Time Frame: predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lomitapide Sprinkled in Applesauce (Treatment A) | Lomitapide Sprinkled in Mashed Banana (Treatment B) | Intact Capsule of 20 mg Lomitapide (Treatment C)
Number analyzed (Participants) | 30 | 30 | 30
ng/mL
  Lomitapide | 0.986 (0.536) | 1.03 (0.463) | 1.13 (0.591)
  M1 | 2.52 (0.748) | 2.65 (0.813) | 2.74 (0.796)
  M3 | 30.2 (15.6) | 31.0 (13.3) | 28.6 (13.7)

3. Primary Outcome: Tmax
Description: Time to reach maximum plasma concentration of lomitapide and its metabolites (M1& M3).
Time Frame: predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Lomitapide Sprinkled in Applesauce (Treatment A) | Lomitapide Sprinkled in Mashed Banana (Treatment B) | Intact Capsule of 20 mg Lomitapide (Treatment C)
Number analyzed (Participants) | 30 | 30 | 30
hours
  Lomitapide | 4.00 [1.00 to 12.0] | 5.00 [1.00 to 12.0] | 5.00 [2.00 to 24.0]
  M1 | 5.00 [2.00 to 8.00] | 5.00 [2.00 to 6.00] | 5.00 [3.00 to 8.00]
  M3 | 2.03 [1.00 to 4.00] | 3.00 [1.00 to 5.00] | 3.00 [1.00 to 4.00]

4. Primary Outcome: t1/2
Description: Terminal elimination half-life of lomitapide and its metabolites (M1& M3).
Time Frame: predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Lomitapide Sprinkled in Applesauce (Treatment A) | Lomitapide Sprinkled in Mashed Banana (Treatment B) | Intact Capsule of 20 mg Lomitapide (Treatment C)
Number analyzed (Participants) | 30 | 30 | 30
h
  Lomitapide | 52.4 (13.3) | 47.7 (12.2) | 48.8 (10.7)
  M1 | 38.7 (7.56) | 37.0 (6.78) | 39.1 (6.32)
  M3 | 46.0 (13.1) | 45.7 (11.5) | 44.0 (11.6)

5. Primary Outcome: AUC0-∞
Description: Area under the plasma concentration vs time curve from zero to infinity of lomitapide and its metabolites (M1& M3).
Time Frame: predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Lomitapide Sprinkled in Applesauce (Treatment A) | Lomitapide Sprinkled in Mashed Banana (Treatment B) | Intact Capsule of 20 mg Lomitapide (Treatment C)
Number analyzed (Participants) | 30 | 30 | 30
ng*h/mL
  Lomitapide | 42.5 (17.7) | 43.8 (15.3) | 47.7 (20.6)
  M1 | 72.8 (20.8) | 75.2 (23.7) | 77.8 (23.9)
  M3 | 457 (317) | 464 (300) | 474 (333)

6. Primary Outcome: λz
Description: Elimination rate constant estimated from individual linear regression of the terminal part of the log concentration vs time curve of lomitapide and its metabolites (M1& M3).
Time Frame: predose and 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 48, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Lomitapide Sprinkled in Applesauce (Treatment A) | Lomitapide Sprinkled in Mashed Banana (Treatment B) | Intact Capsule of 20 mg Lomitapide (Treatment C)
Number analyzed (Participants) | 30 | 30 | 30
1/h
  Lomitapide | 0.0140 (0.00341) | 0.0153 (0.00343) | 0.0149 (0.00320)
  M1 | 0.0185 (0.00344) | 0.0195 (0.00457) | 0.0182 (0.00309)
  M3 | 0.0161 (0.00408) | 0.0162 (0.00428) | 0.0167 (0.00405)

ADVERSE EVENTS:
Arm/Group | Lomitapide Sprinkled in Applesauce (Treatment A) | Lomitapide Sprinkled in Mashed Banana (Treatment B) | Intact Capsule of 20 mg Lomitapide (Treatment C)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 5/30 | 6/31 | 6/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lomitapide Sprinkled in Applesauce (Treatment A) (N=30) | Lomitapide Sprinkled in Mashed Banana (Treatment B) (N=31) | Intact Capsule of 20 mg Lomitapide (Treatment C) (N=31)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Constipation Vomitting
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Described in contract.